CLINICAL TRIAL: NCT02348073
Title: Efficacy of Phosphatidylserine Enriched With Polyunsaturated n-3 Fatty Acid Supplementation on Attention Deficit Disorders in Children With Epilepsy. A Randomized Double-blind Placebo-controlled Trial
Brief Title: Efficacy of Phosphatidylserine Enriched With n-3 PUFA Supplementation on ADHD in Children With Epilepsy
Acronym: AGPIn3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-747
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Last update posted 2025-08-06 (Actual); Status verified 2019-03

CONDITIONS: Attention Deficit Disorder With Hyperactivity; ADHD Inattention or Mixed Type; Epilepsy; Child
Keywords: Epilepsy; Attention Deficit Disorders; VAYARIN; Children; Polyunsaturated n-3 fatty acid supplementation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PS-OMEGA 3, capsules twice daily (Active Comparator): Vayarin®, supplementation of n-3 PUFA: each capsule contains 8.5 mg of docosahexaenoic acid (DHA), 21.5 mg of eicosapentaenoic acid (EPA) and 75 mg of phosphatidylserine.
  Interventions: Drug: Vayarin®, supplementation of n-3 PUFA
- PLACEBO, capsules twice daily (Placebo Comparator): The placebo will be made of cellulose and a small amount of fish powder to maintain the double-blind in odor and taste. The supplementation in n-3 PUFA in the placebo group may be considered as negligible. Placebo will be administered as indistinguishable capsules, identical to the active product.
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: Vayarin®, supplementation of n-3 PUFA — Two capsules will be swallowed twice daily, 20 to 30 minutes prior to breakfast and dinner, during 12 weeks, between visit 1 and visit 2.
  At the end of this period, active product will be continued, at the same dose, for a 12 week-open label period. All patients will be administered the active product.
  Arms: PS-OMEGA 3, capsules twice daily
Drug: PLACEBO — Two capsules will be swallowed twice daily, 20 to 30 minutes prior to breakfast and dinner, during 12 weeks, between visit 1 and visit 2.
  Arms: PLACEBO, capsules twice daily

SUMMARY:
Our project aims to develop a new therapeutic approach in epilepsy-associated attention disorders in children, through evaluation of the clinical impact of dietary n-3 fatty acids, containing eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) conjugated to a phospholipid vector. The primary objective is to evaluate the efficacy of a PUFA supplementation (PS-Omega 3), after 12 weeks of treatment, on attention disorders in children with epilepsy. Secondary objectives include:

* To evaluate the impact of a supplementation of PS-Omega 3 on quality of life.
* To evaluate the impact of a supplementation of PS-Omega 3 on serum and erythrocyte lipid profiles.
* To assess the tolerance of a supplementation of PS-Omega 3.
* To assess the impact of a supplementation of PS-Omega 3 on the frequency of seizures.
* To describe the impact of a supplementation of PS-Omega 3, at 24 weeks,

  1. on attention disorders in children with epilepsy,
  2. on quality of life,
  3. and on serum and erythrocyte lipid profiles. This study will recruit 272 subjects aged 6- 16 years, suffering from epilepsy (any type) and attention deficit hyperactivity disorder (ADHD) (inattentive or combined type) according to DSM V criteria in 12 clinical sites in France.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 15 years and 11 months.
* Children of either sex (male/female) suffering from epilepsy regardless of syndrome classification.
* Subjects on a stable dose of antiepileptic drugs (AED) for at least one month prior to inclusion and subjects for whom no change is considered a priori for the three months following the inclusion.
* Diagnosis of ADHD inattention or mixed type according to the DSM V criteria.
* Subjects must agree to study participation and their parents/legal guardian must provide written inform consent prior to participation in the study.

Exclusion Criteria:

* Subjects less than 6 years or older than 16 years old
* AED not stable for at least one month and/or a change in AED is expected in the three months following inclusion.
* Diagnosis of ADHD hyperactivity type exclusive according to DSM V criteria.
* Mental retardation defined by a score < 70 on the verbal comprehension and perceptual reasoning Wechsler Intelligence Scale for Children - Fourth Edition (WISC-IV), performed within 18 months prior to inclusion or at V1.
* Diagnosis of a psychiatric comorbidity other than ADHD according to the DSM V criteria, including: pervasive developmental disorders including autism disorders; bipolar disordersand psychotic disorders.
* Children suffering from diabetes, any type.
* Use of psychoactive drugs in ADHD within the previous month: Methylphenidate, Amphetamine, Atomoxetine, Modafinil and Antidepressants whatever the class.
* Use of dietary supplementation, other than vitamins, within the last 3 months.
* Use of ketogenic diet within the last 3 months.
* Allergy to fish or other sea products.
* Soy allergy.
* Absence of coverage by social security.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Reduction of the ADHD-rating scale IV inattentive subscore in subjects assigned to supplementation of PS-Omega 3 in comparison with the placebo group after 12 weeks of treatment. | 12 weeks
  The ADHD Rating Scale-IV quantifies each of the 18 symptoms of ADHD on a 0 to 3 scale, with a maximum score of 54 points. Nine of the 18 items score for inattention while the nine others assess hyperactivity with a maximum of 27 points each. The discriminative value of these two subscales was validated, allowing their individual use.

SECONDARY OUTCOMES:
Reduction of the ADHD Rating Scale-IV total score in the PS-Omega 3 group compared with the placebo group after 12 weeks of treatment. | 12 weeks
  The ADHD Rating Scale-IV quantifies each of the 18 symptoms of ADHD on a 0 to 3 scale, with a maximum score of 54 points.
Reduction of TOVA total score in the PS-Omega 3 group compared with the placebo group after 12 weeks of treatment. | 12 weeks
  The TOVA (Test of Variables of Attention) is a computerized tool assessing the capacity of attention and impulse control. This test has been validated as a diagnostic tool in ADHD.
Proportion of subjects with a normalized TOVA score in the PS-Omega 3 group compared with the placebo group after 12 weeks of treatment. | 12 weeks
  The TOVA (Test of Variables of Attention) is a computerized tool assessing the capacity of attention and impulse control. This test has been validated as a diagnostic tool in ADHD.
Change in quality of life score in the PS-Omega 3 group compared with the placebo group after 12 weeks of treatment. | 12 weeks
  Quality of life assessed by the EFIQUACEE questionnaire (Echelle Française d'Impact et de Qualité de Vie Chez l'Enfant atteint d'Epilepsie).
  The EFIQUACEE questionnaire is a unique quality of life scale for children suffering from epilepsy. It is validated in French language.
Evolution of plasma lipid profiles in subjects assigned to supplementation of PS-Omega 3 in comparison with the placebo group after 12 weeks of treatment. | 12 weeks
  Plasma levels before and after 12 weeks of treatment: total lipid mass ; total phospholipids ; individual phospholipids including: lysophosphatidylcholin, phosphatidylcholin, sphingomyelin, phosphatidylserine, phosphatidylinositol, phosphatidylethanolamine, diphosphatidylglycerol, lysophosphatidylethanolamine ; total triglycerides ; fatty acids profiles in phospholipids; fatty acids profiles in triglycerides ; fatty acids profiles in cholesterol esters.
Evolution of eythrocytes lipid profiles in subjects assigned to supplementation of PS-Omega 3 in comparison with the placebo group after 12 weeks of treatment. | 12 weeks
  Quantification of, in erythrocyte membrane, before and after 12 weeks of treatment: total lipid mass ; total phospholipids ; individual phospholipids including: lysophosphatidylcholin, phosphatidylcholin, sphingomyelin, phosphatidylserine, phosphatidylinositol, phosphatidylethanolamine, diphosphatidylglycerol, lysophosphatidylethanolamine ; total triglycerides ; fatty acids profiles in phospholipids; fatty acids profiles in triglycerides ; fatty acids profiles in cholesterol esters.
Tolerance of a supplementation of PS-Omega 3. | 36 weeks
  Tolerance analysis of the supplementation of PS-Omega 3: interrogatoire, phone calls, clinical examinations, adverse events reported throughout the study.
Number of subjects with a reduction in the frequency of seizures ≥ 50%, in the PS-Omega 3 group compared with the placebo group after 12 weeks of treatment. | 12 weeks
After 24 weeks of treatment, description of the total score of ADHD Rating Scale. | 24 weeks
After 24 weeks of treatment, description of the total score of TOVA. | 24 weeks
After 24 weeks of treatment, proportion of subjects with a normalized TOVA score. | 24 weeks
After 24 weeks of treatment, change in quality of life score (EFIQUACEE questionnaire). | 24 weeks
After 24 weeks of treatment, plasma lipid levels before and after treatment. | 24 weeks
  Plasma levels before and after 24 weeks of treatment: total lipid mass ; total phospholipids ; individual phospholipids including: lysophosphatidylcholin, phosphatidylcholin, sphingomyelin, phosphatidylserine, phosphatidylinositol, phosphatidylethanolamine, diphosphatidylglycerol, lysophosphatidylethanolamine ; total triglycerides ; fatty acids profiles in phospholipids; fatty acids profiles in triglycerides ; fatty acids profiles in cholesterol esters.
After 24 weeks of treatment, erythrocyte lipid levels before and after treatment. | 24 weeks
  Quantification of, in erythrocyte membrane, before and after 24 weeks of treatment: total lipid mass ; total phospholipids ; individual phospholipids including: lysophosphatidylcholin, phosphatidylcholin, sphingomyelin, phosphatidylserine, phosphatidylinositol, phosphatidylethanolamine, diphosphatidylglycerol, lysophosphatidylethanolamine ; total triglycerides ; fatty acids profiles in phospholipids; fatty acids profiles in triglycerides ; fatty acids profiles in cholesterol esters.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Rheims, MD, Principal Investigator — Hospices Civils de Lyon
Locations (13):
- France (13):
  - CHU de Amiens, Amiens
  - CHU d'Angers, Angers
  - Hôpital des Enfants - Pellegrin, Bordeaux
  - CHRU Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - Hôpital de la Timone, Marseille
  - Hôpital Necker-Enfants malades, Paris
  - Hôpital Robert-Debré, Paris
  - CHU de Rennes, Rennes
  - Hôpital de Hautepierre, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHU de Tours, Tours
  - Hôpital Brabois - Rue du Morvan, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Rheims S, Herbillon V, Gaillard S, Mercier C, Villeuve N, Villega F, Cances C, Castelnau P, Napuri S, de Saint-Martin A, Auvin S, Nguyen The Tich S, Berquin P, de Bellecize J, Milh M, Roy P, Arzimanoglou A, Bodennec J, Bezin L, Kassai B; investigators of the AGPI study group. Phosphatidylserine enriched with polyunsaturated n-3 fatty acid supplementation for attention-deficit hyperactivity disorder in children and adolescents with epilepsy: A randomized placebo-controlled trial. Epilepsia Open. 2024 Apr;9(2):582-591. doi: 10.1002/epi4.12892. Epub 2024 Jan 25. PMID 38173190
- [Derived] Gillies D, Leach MJ, Perez Algorta G. Polyunsaturated fatty acids (PUFA) for attention deficit hyperactivity disorder (ADHD) in children and adolescents. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD007986. doi: 10.1002/14651858.CD007986.pub3. PMID 37058600